CLINICAL TRIAL: NCT02448329
Title: Study of AZD1775 in Combination With Paclitaxel, in Advanced Gastric Adenocarcinoma Patients Harboring TP53 Mutation as a Second-line Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-04-127
Record Dates: First submitted 2015-05-13; First posted 2015-05-19 (Estimated); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Advanced Gastric Adenocarcinoma
MeSH Terms: interventions — adavosertib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD1775 in Combination With Paclitaxel (Experimental): AZD1775 225 mg BID q 12 hours (x 5 doses, 2.5 days) administered days 1~3 Weekly paclitaxel 80 mg/m2 IV on 1, 8 and 15 of a four week l cycle is an widely used dose of paclitaxel given on this schedule in gastric adenocarcinoma patients as second-line therapy.
  Interventions: Drug: AZD1775; Drug: paclitaxel

INTERVENTIONS:
Drug: AZD1775 — AZD1775 225 mg BID q 12 hours (x5 doses, 2.5 days) administered days 1~3
Drug: paclitaxel — paclitaxel 80 mg/m2 given days 1, 8 and 15 of a 28 day cycle

SUMMARY:
This study is a single arm, single center phase II study of AZD1775 in combination with paclitaxel in patients with advanced gastric adenocarcinoma harboring TP53 mutation as a second-line chemotherapy.

Patients will receive AZD 1775 plus weekly paclitaxel combination regimen. The arm is composed of 25 patients.

AZD1775 225 mg BID q 12 hours (x 5 doses) administered days 1~3 + paclitaxel 80 mg/m2 given days 1, 8 and 15 of a 28 day cycle.

Tumour evaluation using Response Evaluation Criteria in Solid Tumors 1.1 will be conducted at screening every 16 weeks until objective disease progression .

DETAILED DESCRIPTION:
AZD1775 is an inhibitor of Wee1, a protein tyrosine kinase. Wee1 phosphorylates and inhibits cyclin-dependent kinases 1 (CDK1) and 2 (CDK2), and is involved in regulation of the intra-S and G2 cell cycle checkpoints.

In in vitro and in vivo preclinical models, AZD1775 selectively enhanced chemotherapy induced death of cells deficient in p53 signaling. Tumor context-specific sensitization to the DNA damaging agents gemcitabine and platinums was observed in TOV21G (ovarian carcinoma) cell lines matched for wild type and knock down of p53.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥20 years of age.
3. Advanced gastric adenocarcinoma (including GEJ) that has progressed during or after first line therapy.

   * The 1st line regimen must have contained doublet 5-fluoropyrimidine or platinum based regimen.
   * Relapse within 6 months of completion of adjuvant/neoadjuvant chemotherapy containing doublet 5-fluoropyrimidine and platinum-based regimen could be considered as 1st line therapy.
4. Previous adjuvant/neoadjuvant chemotherapy is allowed, if completed more than 6 months prior to starting the 1st line therapy.
5. Provision of tumor sample (from either a resection or biopsy)
6. Patients with p53mutation
7. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
8. Eastern Cooperative Oncology Group performance status 0-1
9. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
10. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥9.0 g/dL (transfusion allowed)
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * White blood cells (WBC) > 3 x 109/L
    * Platelet count ≥100 x 109/L (transfusion allowed)
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
    * aspartate aminotransferase (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
    * Serum creatinine ≤1.5 x institutional ULN
11. At least one measurable lesion that can be accurately assessed by imaging or physical examination at baseline and following up visits.
12. Negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1.

Exclusion Criteria:

1. More than one prior chemotherapy regimen (except for adjuvant/neoadjuvant chemotherapy with more than 6 month wash out period) for the treatment of gastric cancer in the advanced setting.
2. Any previous treatment with P53 inhibitors (small molecules)
3. Any previous treatment with paclitaxel
4. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer,curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≤5 years.
5. HER2 positive patients (defined by HER2 3+ by immunohistochemistry or HER2 SISH +)
6. Patients unable to swallow orally administered medication.
7. Treatment with any investigational product during the last 14 days before the enrollment (or a longer period depending on the defined characteristics of the agents used).
8. Patients receiving any systemic chemotherapy, radiotherapy (except for palliative reasons), within 3 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used). The patient can receive a stable dose of bisphosphonates or denusomab for bone metastases, before and during the study as long as these were started at least 4 weeks prior to treatment.
9. Concomitant use of known potent CYP3A4 inhibitors such as ketoconazole, itraconazole,ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir.
10. With the exception of alopecia, any ongoing toxicities (>Common Toxicity Criteria for Adverse Effects grade 1) caused by previous cancer therapy.
11. Intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
12. Resting ECG with measurable QTcB > 480 msec on 2 or more time points within a 24hour period or family history of long QT syndrome.
13. Patients with cardiac problem as follows: uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy) Left ventricular ejection fraction <55% measured by echocardiography, Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest , Symptomatic heart failure (NYHA grade II-IV), Prior or current cardiomyopathy, Severe valvular heart disease, Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy), Acute coronary syndrome within 6 months prior to starting treatment
14. Ophthalmological conditions as follows:Intra-ocular pressure >21 mmHg, or uncontrolled glaucoma (irrespective of intra-ocular pressure), Current or past history of central serous retinopathy or retinal vein occlusion
15. Female patients who are breast-feeding or child-bearing
16. Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV)

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 8weeks

SECONDARY OUTCOMES:
Duration of response | 24weeks
Disease control rate | 8weeks
Overall survival | 24weeks
progression-free survival (PFS) | 24weeks
safety and tolerability measured by Adverse Events,Vital signs,Collection of clinical chemistry/haematology parameters,ECGs | 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jee yun Lee, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical center, Seoul, South Korea